CLINICAL TRIAL: NCT03457337
Title: A Randomized, Controlled, Open-label, Prospective Trial of S-1 Plus Gefitinib Versus Gefitinib Monotherapy for First-line Treatment of Advanced Non-squamous Non-small Cell Lung Cancer With EGFR-sensitive Mutation
Brief Title: S-1 Plus Gefitinib Versus Gefitinib Monotherapy in Patients With EGFR-sensitive Mutation Advanced Non-squamous NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA-01
Record Dates: First submitted 2018-02-23; First posted 2018-03-07 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-04

CONDITIONS: Advanced NSCLC With EGFR Mutation
MeSH Terms: interventions — S 1 (combination); Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-1 plus Gefitinib (Experimental): S-1: According to the body surface area (BSA) to determine the dose, twice daily, after breakfast and dinner orally, continuous administration of 14 days, rest for 7 days. BSA <1.25 m2, 80 mg / day; BSA 1.25 m2 to <1.5 m2, 100 mg / day; BSA 1.5 m2 or more, 120 mg / day. Until disease progression, intolerance of toxicity or withdrawal of informed consent from the subject.
  Gefitinib: 250mg, 1 day, orally, fasting or with the same service. Until disease progression, intolerance of toxicity or withdrawal of informed consent from the subject.
  Interventions: Drug: S-1 plus Gefitinib
- Gefitinib (Active Comparator): Gefitinib 250 mg/day oral daily
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: S-1 plus Gefitinib — S-1: According to the body surface area (BSA) to determine the dose, twice daily, after breakfast and dinner orally Gefitinib: 250mg, 1 day, orally, fasting or with the same service
  Arms: S-1 plus Gefitinib
Drug: Gefitinib — Gefitinib: 250mg, 1 day, orally
  Arms: Gefitinib

SUMMARY:
To investigate the survival benefit of first-line therapy for patients with EGFR-sensitive mutation-positive advanced non-squamous non-small cell lung cancer treated with S-1plus gefitinib versus gefitinib monotherapy

DETAILED DESCRIPTION:
This is a randomized, controlled, open-plan, prospective clinical study. According to the available evidence, we selected patients with locally advanced or metastatic non-squamous non-small cell lung cancer with stage Ⅲ-C-Ⅳ confirmed by cytology or histology and positive EGFR-sensitive mutation, then patients accept first-line treatment with S-1 plus gefitinib or gefitinib. This study will collect FFS during treatment until the patient dies and will follow the survival of the subject after the disease progresses.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteered for attending the study, and signed informed consent form (ICF)to participate in the study.
2. Males or females aged ≥18 years, < 75 years.
3. Cytologically and Histologically documented, advanced or recurrent (stage IIIc-IV) non-small cell lung cancer patients .
4. exon 19 deletion or exon 21 L858R for EGFR mutation.
5. Patients hadn't received past system treatment, including cytotoxic drugs; For patients who have received adjuvant or neoadjuvant chemotherapy appears recurrence or metastasis more than 6 months from accepting the last dose of chemotherapy drugs
6. Patients must have at least 1 measurable lesion according to the RECIST (version 1.1) criteria.
7. Life expectancy ≥12 weeks.
8. ECOG performance status 0-2.
9. Adequate organ function as defined by the following criteria:

   Absolute neutrophil count (ANC) ≥1.5 x 109/L, and Platelet count ≥100 x 109/L, and Hemoglobin ≥9 g/dL (may be transfused to maintain or exceed this level).

   Total bilirubin ≤ 1.5 x upper limit of normal (ULN), alkaline phosphatase (AP), Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x ULN in the absence of liver metastases or up to 5 ULN in case of liver metastases.

   creatinine clearance≥ 60 ml/min.
10. Fertile men and women must use effective contraception.
11. Subjects are allowed to receive radiation for lesions other than the target lesion, but the end of radiotherapy should be at least 3 weeks apart from randomization;
12. The investigators should judge the subject's compliance to meet the study requirements.

Exclusion Criteria:

1. Histology confirmed for squamous carcinomas, including mixed gland scale cancer, small cell lung cancer.
2. Patients with prior any anti-tumor therapy,including chemotherapy, radiotherapy, immunotherapy or biotherapy
3. Patients with prior exposure to EGFR-TKIs or 5-Fu
4. Not recovered from previous toxic reactions for anticancer treatment (CTCAE grade 1) or not fully recovered from previous surgery
5. Patients who have brain metastasis. It is permitted if the patient has been treated with surgery and/or radiation with evidence of stable disease for at least 4 weeks.
6. Patients haven't been diagnosed other malignant disease, except the basal cell carcinoma and cervical carcinoma.
7. A uncontrolled clinical infection, activity, including acute pneumonia,HIV,HCV. , etc.
8. Sullivudine, brivudine or other antiviral drugs of similar structure were used within 2 months before randomization
9. Patients who have a difficulty in swallowing or drug absorption.
10. Patients with a history of interstitial lung disease or with interstitial lung disease;
11. There are diseases of alimentary canal such as active duodenal ulcer, the ulcerous colitis, intestinal obstruction or other conditions which can cause gastrointestinal bleeding or perforation in the investigator's opinion; or patient has a history of intestinal perforation, intestinal fistula.
12. Evaluation of cardiac function: left ventricular ejection fraction < 50% (echocardiography); Moderate or above disorders of mitral valve and tricuspid shut down;, serious/unstable angina or acute myocardial infarction coronary artery bypass surgery in 6 months before enrollment; patients with class 2 and above cardiac dysfunction according to New York heart association (NYHA) classification
13. Patients with medical history of hemoptysis (defined as about 2.5ml bright blood) 2 weeks before the enrollments
14. Stroke and transient ischemic in 12 months before enrollment.
15. Severe ulcer in the skin wound, trauma and mucosa or fractures have been not fully healed.
16. Patients received CYP3A4 strong inhibitor and/or inducer in 2 weeks before enrollment; Patients received P-gp and breast cancer resistance protein (BCRP) substrates drug in 2 weeks before enrollment.
17. Patients has participated in other clinical trials of antitumor drugs within the previous 28 days, except for those who were able to prove that they were using placebo;
18. Pregnancy or lactating women or pregnant women may be pregnant before pregnancy test positive;
19. Unwillingness to receive contraception by patients or their sexual partners who are fertile but unwilling to receive contraception;
20. The investigators think that there is any clinical or laboratory abnormalities in the subjects that are not suitable for this study.
21. There is a serious psychological or mental abnormalities, researchers assess subjects to participate in this clinical study compliance is insufficient;
22. Allergic reactions to analogs of gefitinib and S-1 and / or Analogs and / or excipients in test drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) | 2 years
  From start of anti-cancer therapy until progression or death.To evaluate the disease free survival of gefitinib combined with S-1 and gefitinib in patients with Pathological stage IIIc-IV NSCLC harbouring sensitive mutations of EGFR. Progression free survival (PFS)- defined as the time from initial medication to the first documented disease progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  To evaluate the overall survivalof gefitinib combined with S-1 and gefitinib in patients with Pathological stage IIIc-IV NSCLC harbouring sensitive mutations of EGFR in the 3 years since treatment begain
Disease control rate | 2 years
  To compare disease control rate of the two arms from start of anti-cancer therapy until progression
Objective response rate(ORR) | 2 years
  To compare objective response rate of the two arms from start of anti-cancer therapy until progression
Number of Participants with Adverse Events | 3 years
  The safety and tolerability profile of gefitinib at a 250 mg daily dose relative to that of radiotherapy.

OTHER OUTCOMES:
Assessment of Health-related quality of life | 3 years
  Quality of Life Questionnaire(such as QLQ-C30 and QLQ-LC13) evaluated since treatment began.At the end of the trial, the differences between the two indicators were compared with Mixed-effects model repeated measures (MMRM), where the baseline was scored as a covariant and the treatment group as a fixed variable. In addition, the baseline values of the two scores, the value of each visit, and the change value of the baseline were statistically described.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China